CLINICAL TRIAL: NCT00512174
Title: Prospective Trial to Evaluate Efficacy and Accuracy of a Portable Ultrasound Scanner for Non-Invasive Bladder Volume Measurement (BladderScan BVI3000) in Patients After Radical Cystectomy and Bladder Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHEBA-07-4629-ZD-CTIL
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2007-08-07 (Estimated); Status verified 2007-08

CONDITIONS: Bladder Substitution; Reconstructed Bladder
Keywords: Portable Ultrasound Scanner; Non Invasive Bladder Volume Measurement; Radical Cystectomy; Bladder Reconstruction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: BladderScan BVI 3000

SUMMARY:
Thirty patients who underwent radical cystectomy and bladder substitution and thirty people with native bladders will be enrolled in the study. After meticulous explanations each person will undergo sterile catheterization of the bladder/neobladder with a 14 Fr Foley catheter. After catheterization the bladder will be fully emptied. Randomly assigned volume of sterile saline will be injected to the bladder via the catheter by one sub investigator and the bladder capacity will be measured via a portable ultrasound scanner for non-invasive bladder volume measurement (BladderScan BVI3000) by another sub investigator. The volume injected and the measured results will remain in a closed envelope till the completion of the trial. After each measurement the first sub investigator will completely empty the bladder/neobladder and the process will repeat itself for a total of six measurements for each patient or first mention of discomfort (whichever comes first), after which the bladder will be drained once more and the catheter removed.

ELIGIBILITY:
Inclusion Criteria:

Group A: Patients ages 18-75, at least 6 month after radical cystectomy and bladder substituition Group B: Volunteers same age group as group A, with native bladder as control group

Exclusion Criteria:

Group A: carrying ureteral stent of any kind, inability to catheterize patient due to severe urethral stricture, incarcerated post operative ventral hernia, after mesh repair of POVH, active urinary tract infection, acute bacterial prostatitis.

Group B: patients after partial cystectomy, incarcerated post operative ventral hernia, after mesh repair of POVH, active urinary tract infection, acute bacterial prostatitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-08

PRIMARY OUTCOMES:
Efficacy and Accuracy of a Portable Ultrasound Scanner for Non-Invasive Bladder Volume Measurement (BladderScan BVI3000) in Patients After Radical Cystectomy and Bladder Reconstruction | 12 Month

CONTACTS AND LOCATIONS:
Overall Officials: Zohar Dotan, M.D, PhD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Byun SS, Kim HH, Lee E, Paick JS, Kamg W, Oh SJ. Accuracy of bladder volume determinations by ultrasonography: are they accurate over entire bladder volume range? Urology. 2003 Oct;62(4):656-60. doi: 10.1016/s0090-4295(03)00559-4. PMID 14550437